CLINICAL TRIAL: NCT05501054
Title: Phase 1b/2 Trial of Ipilimumab, Nivolumab, and Ciforadenant (Adenosine A2a Receptor Antagonist) in First-line Advanced Renal Cell Carcinoma.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0093; NCI-2022-06736 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ipilimumab; Nivolumab; ciforadenant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipilimumab, Nivolumab, and Ciforadenant (Experimental): To help control advanced renal cell carcinoma.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Ciforadenant

INTERVENTIONS:
Drug: Ipilimumab — Given by IV (vein)
  Other Names: Yervoy; BMS-734016; MDX010
Drug: Nivolumab — Given by IV (vein)
  Other Names: BMS-936558; Opdivo
Drug: Ciforadenant — Given by PO

SUMMARY:
To learn if the combination of ciforadenant, ipilimumab, and nivolumab can help to control advanced renal cell carcinoma

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the safety and tolerability of ipilimumab, nivolumab, and ciforadenant in patients with untreated advanced renal cell carcinoma (RCC).
* To assess the depth of responsein patients with untreated advanced renal cell carcinoma treated with ipilimumab, nivolumab, and ciforadenant.

Secondary Objectives:

• To estimate the objective response rate (ORR), duration of response (DOR) progression free survival (PFS), progressive disease (PD) rate, and irAE rate of ipilimumab, niovlumab, and Ciforadenant combination in untreated advanced RCC.

Exploratory Objectives:

• To assess association of gene expression signatures and pharmacodynamic parameters with outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Willing and able to provide a signed and dated written informed consent
2. Male or female ≥ 18 years of age
3. Confirmed diagnosis of clear cell RCC
4. Stage IV metastatic renal cell carcinoma per American Joint Committee on Cancer
5. No prior systemic therapy for advanced RCC
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 2)
7. At least one measureable lesion as defined by RECIST 1.1

   • A tumor lesion situated in a previously irradiated area is considered a measureable/target lesion only if subsequent disease progression has been documented in the lesion
8. Has submitted an archival tumor tissue sample or newly obtained core or incisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed parrafin-embedded tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue but not necessary. Details pertaining to tumor tissue submission can be found in the Lab Procedures Manual
9. Willing and able to under go bone and brain scans at baseline and continue to have scans performed if positive at screening.
10. Adequate organ function within 21 days prior to first dose of protocol-indicated treatment, including:

    * White blood cell (WBC) ≥ 2,000 /µL
    * Absolute neutrophil count (ANC) ≥ 1,500/µL
    * Platelets ≥ 100,000/µL
    * Hemoglobin (Hgb) ≥ 9.0 g/d without requirement for transfusion in prior 4 weeks
    * Serum creatinine ≤ 2 times institutional upper limit of normal (ULN), or calculated creatinine clearance ≥ 40 mL/min (per the Cockcroft-Gault formula, Appendix 3)
    * Total bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who must have total bilirubin < 3.0 mg/dL)
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
11. Women must not be breastfeeding while taking the study drug and for up to five months after the last dose of study drug
12. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to receiving first dose of protocol-indicated treatment

    * "Women of childbearing potential" (WOCBP) is defined as any female who has experienced menarche who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal
    * Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 years of age in the absence of other biological or physiological causes
    * If menopausal status is considered for the purpose of evaluating childbearing potential, women < 62 years of age must have a documented serum follicle stimulating hormone (FSH) level within laboratory reference range for postmenopausal women, in order to be considered postmenopausal and not of childbearing potential
13. Women of childbearing potential (WOCBP) must agree to follow instructions for acceptable contraception Appendix 4 from the time of signing consent, and for 23 weeks after their last dose of protocol-indicated treatment
14. Men not azoospermic who are sexually active with WOCBP must agree to follow instructions for acceptable contraception (Appendix 4), from the time of signing consent, and for 31 weeks after their last dose of protocol-indicated treatment

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from the trial:

1. Prior systemic treatment including neoadjuvant or adjuvant therapy <6 months from protocol initiation is not allowed including an immune checkpoint inhibitor or TKI
2. ≤ 28 days before first dose of protocol-indicated treatment:

   * Major surgery requiring general anesthesia
   * Suspected or confirmed SARS-CoV-2 infection
3. ≤ 14 days before first dose of protocol-indicated treatment:

   * Radiosurgery or radiotherapy
   * Minor surgery. (Note: Placement of a vascular access device is not considered minor or major surgery)
   * Active infection requiring infusional treatment
4. Known or suspected clinically significant active bleeding including active hemoptysis
5. Inability to swallow oral medication; or the presence of a poorly controlled gastrointestinal disorder that could significantly affect the absorption of oral study drug - e.g. Crohn's disease, ulcerative colitis, chronic diarrhea (defined as > 4 loose stools per day), malabsorption, or bowel obstruction
6. Central nervous system (CNS) metastasis, unless asymptomatic and stable with imaging of the head by MRI unless contraindicated for the patient in which case CT is acceptable showing no change in CNS disease status for at least two (2) weeks prior to initiating protocol-indicated treatment
7. Any condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone or equivalent daily) or other immunosuppressive medications within 14 days prior to initiating protocol-indicated treatment

   • In the absence of active autoimmune disease: Subjects are permitted the use of corticosteroids with minimal systemic absorption (e.g. topical, ocular, intra-articular, intranasal, and inhalational) ≤ 10 mg/day prednisone or equivalent daily; and physiologic replacement doses of systemic corticosteroids ≤ 10 mg/day prednisone or equivalent daily (e.g. hormone replacement therapy needed in patients with hypophysitis)
8. Active, known or suspected autoimmune disease

   • Subjects with type I diabetes mellitus; hypothyroidism only requiring hormone replacement; skin disorders such as vitiligo, psoriasis or alopecia not requiring systemic treatment; or conditions not expected by the investigator to recur in the absence of an external trigger are permitted to enroll
9. Known psychiatric condition, social circumstance, or other medical condition reasonably judged by the investigator to unacceptably increase the risk of study participation; or to prohibit the understanding or rendering of informed consent or anticipated compliance with and interpretation of scheduled visits, treatment schedule, laboratory tests and other study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
To establish the objective response rate (ORR) | through study completion and average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Duke Cancer Institute, Durham, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org